CLINICAL TRIAL: NCT02358681
Title: Intranasal Ketorolac Versus Intravenous Ketorolac for Treatment of Migraine Headaches in Children: A Randomized Non-inferiority Clinical Trial
Brief Title: Intranasal Ketorolac Versus Intravenous Ketorolac for Treatment of Migraine Headaches in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Migraine Research Foundation (Other)
Responsible Party: Principal Investigator, Daniel S Tsze, MD, MPH, Assistant Professor of Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAO1302
Record Dates: First submitted 2015-01-29; First posted 2015-02-09 (Estimated); Results first posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Migraine
Keywords: Intranasal; Ketorolac; Pediatric; Migraine; Headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketorolac, intranasal (Experimental): 1. Ketorolac 1 mg/kg, maximum dose 30 mg. To be administered by intranasal route, single dose.
  2. Placebo, intravenous.
  Interventions: Drug: Ketorolac, intranasal; Drug: Placebo, intravenous
- Ketorolac, intravenous (Active Comparator): 1. Ketorolac 0.5 mg/kg, maximum dose 30 mg. To be administered by intravenous route, single dose.
  2. Placebo, intranasal.
  Interventions: Drug: Ketorolac, intravenous; Drug: Placebo, intranasal

INTERVENTIONS:
Drug: Ketorolac, intranasal — Ketorolac 1 mg/kg, maximum dose 30 mg. To be administered by intranasal route.
  Other Names: Toradol
  Arms: Ketorolac, intranasal
Drug: Ketorolac, intravenous — Ketorolac 0.5 mg/kg, maximum dose 30 mg. To be administered by intravenous route.
  Other Names: Toradol
  Arms: Ketorolac, intravenous
Drug: Placebo, intravenous — Placebo of equal volume to IV ketorolac, to be administered by intravenous route.
  Arms: Ketorolac, intranasal
Drug: Placebo, intranasal — Placebo of equal volume to IN ketorolac, to be administered by intranasal route.
  Arms: Ketorolac, intravenous

SUMMARY:
Ketorolac is an evidence-based, first-line acute migraine therapy that is commonly used in the pediatric population; however, it is typically administered by the intravenous (IV) or intramuscular (IM) routes, both of which require a painful and distressing needle stick to administer.

The intranasal (IN) route is a painless and effective way of administering analgesics, including ketorolac: IN ketorolac has been shown to be an effective analgesic in adults for painful conditions, including acute migraine headaches. However, IN ketorolac has been understudied in children, and it is not known how effective it is compared to IV ketorolac, which is currently the most common way of administering ketorolac to children. If IN ketorolac is shown to be no less effective than IV ketorolac, IN ketorolac may be a viable and painless alternative to effectively treat acute migraine headaches in children.

Therefore, our primary aim is to demonstrate that IN ketorolac is non-inferior to IV ketorolac for reducing pain in children with acute migraine headaches.

DETAILED DESCRIPTION:
Primary Aim: Determine whether intranasal (IN) ketorolac is non-inferior to intravenous (IV) ketorolac for reducing pain in children with acute migraine headaches. We hypothesize that IN ketorolac is non-inferior to IV ketorolac in reducing acute migraine headache pain by a minimum clinically significant difference within 60 minutes of administration.

Secondary Aim: Determine whether there is a difference in time to achieve a clinically significant reduction in pain after receiving IN ketorolac compared to IV ketorolac. We hypothesize that there is no difference between IN ketorolac and IV ketorolac in the time it takes to achieve a clinically significant reduction in pain.

We will conduct a prospective, double-blinded, randomized, non-inferiority, parallel 1:1 clinical trial of eligible children in a single urban pediatric ED. We will block randomize patients to receive either 1 mg/kg IN ketorolac and an IV placebo (study group A), or 0.5 mg/kg IV ketorolac and an IN placebo (study group B).

We will assess the patient's pain at baseline, and then at 10 minutes, 30 minutes and 60 minutes after administration of the study drug. The patient will then be assessed at 2 hours and 24 hours after study drug administration for outcomes related to efficacy, function, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Present to the emergency department with a migraine headache as defined by the modified Irma criteria. The modified Irma criteria are as follows: Headache episodes of 1-168 hours (7 days) presenting with at least 3 of the following 6 criteria: moderate to severe episode of impaired daily activities; focal localization of headache; pulsatile description; nausea or vomiting or abdominal pain; photophobia or phonophobia or avoidance of light and noise; symptoms increasing with activity or resolving by rest.
* Headache severity of moderate to severe pain (i.e. at least 4/10 on the Faces Pain Scale - Revised)
* Requiring IV fluids and any IV medication (for example: ketorolac, metoclopramide, prochlorperazine, ondansetron) as part of their headache treatment, as per their treating attending physician

Exclusion Criteria:

* Contraindication to receiving ketorolac
* Receipt of an NSAID within six hours of study drug administration
* Presence of an intranasal obstruction that cannot be readily cleared
* Inability to speak English or Spanish
* Unable to complete self-report measures of pain or questionnaires
* Critical illness
* Frequent use of drugs for headache (i.e. regular intake of analgesics for acute headaches on more than 10 days per month).

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Tsze, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- NewYork Presbyterian Morgan Stanley Children's Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketorolac, Intranasal: 1. Ketorolac 1 mg/kg, maximum dose 30 mg. To be administered by intranasal route, single dose.
  2. Placebo, intravenous.
  Ketorolac, intranasal: Ketorolac 1 mg/kg, maximum dose 30 mg. To be administered by intranasal route.
  Placebo, intravenous: Placebo of equal volume to IV ketorolac, to be administered by intravenous route.
- Ketorolac, Intravenous: 1. Ketorolac 0.5 mg/kg, maximum dose 30 mg. To be administered by intravenous route, single dose.
  2. Placebo, intranasal.
  Ketorolac, intravenous: Ketorolac 0.5 mg/kg, maximum dose 30 mg. To be administered by intravenous route.
  Placebo, intranasal: Placebo of equal volume to IN ketorolac, to be administered by intranasal route.
Period: Overall Study
Arm/Group | Ketorolac, Intranasal | Ketorolac, Intravenous
Started | 29 | 30
Completed | 27 | 29
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac, Intranasal | Ketorolac, Intravenous | Total
Number analyzed (Participants) | 27 | 29 | 56
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14 [11 to 16] | 15 [11 to 16] | 14.5 [11 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 10 | 8 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 24 | 26 | 50
  Black | 2 | 0 | 2
  White | 0 | 3 | 3
  Don't know | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score After Analgesic Administration (Faces Pain Scale - Revised (FPS-R)
Description: Measure the change in pain score after administration of analgesic using the Faces Pain Scale - Revised (FPS-R) at 60 minutes after analgesic administration. The FPS-R is scored from 0 (no pain) to 10 (maximum pain intensity, i.e. worst outcome).
Time Frame: 60 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ketorolac, Intranasal | Ketorolac, Intravenous
Number analyzed (Participants) | 27 | 29
units on a scale | 4.2 [3.6 to 4.8] | 4.4 [3.5 to 5.3]

2. Secondary Outcome: Time to Achieve Clinically Significant Reduction in Pain After Analgesic Administration (Pain Score)
Description: Pain score will be assessed at 10, 30, 60 and 120 minutes after analgesic administration, until pain score decreases by 2/10 on the Faces Pain Scale - Revised (FPS-R). The FPS-R is scored from 0 (no pain) to 10 (maximal pain, i.e. worst outcome)
Time Frame: 10, 30, 60 and 120 minutes
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Ketorolac, Intranasal | Ketorolac, Intravenous
Number analyzed (Participants) | 27 | 29
Minutes | 21.9 [15 to 28.8] | 18.6 [12.7 to 25]

3. Other Pre Specified Outcome: Adverse Events
Description: Adverse events will be assessed at the 1- and 2-hour assessments and the 24-hour follow up.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac, Intranasal | Ketorolac, Intravenous
Number analyzed (Participants) | 27 | 29
Participants | 0 | 1

4. Other Pre Specified Outcome: Number of Participants Who Received Rescue Medications During Emergency Department Visit
Description: Rescue medication defined as an additional parenteral analgesic administered in response to inadequate improvement in pain. Rescue medication was administered when deemed clinically indicated by the treating clinician.
Time Frame: 12 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac, Intranasal | Ketorolac, Intravenous
Number analyzed (Participants) | 27 | 29
Participants | 6 | 5

5. Other Pre Specified Outcome: Number of Participants Who Experienced Headache Relief During Emergency Department Visit
Description: Headache relief defined as change of the patient's headache pain intensity from severe to moderate to either mild or none, without receipt of rescue medications.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac, Intranasal | Ketorolac, Intravenous
Number analyzed (Participants) | 27 | 29
Participants | 25 | 26

6. Other Pre Specified Outcome: Number of Participants Who Experienced Headache Freedom During Emergency Department Visit
Description: Headache freedom defined as achieving a headache pain intensity of "none", without receipt of rescue medications.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac, Intranasal | Ketorolac, Intravenous
Number analyzed (Participants) | 27 | 29
Participants | 11 | 17

7. Other Pre Specified Outcome: Percentage Change in Pain Score Between Baseline and One Hour
Description: Percentage change in pain score between baseline and one hour after study medication administration. Pain measured using the Faces Pain Scale - Revised (FPS-R), which is scored from 0 (no pain) to 10 (maximum pain intensity, i.e. worst outcome). Positive values (i.e. percentage change) indicate a DECREASE (i.e. improvement) in pain intensity.
Time Frame: 1 hour
Measure: Mean (95% Confidence Interval); unit: percentage of initial pain intensity
Arm/Group | Ketorolac, Intranasal | Ketorolac, Intravenous
Number analyzed (Participants) | 27 | 29
percentage of initial pain intensity | 69.8 [60.6 to 78.9] | 71.8 [60.7 to 82.9]

8. Other Pre Specified Outcome: Number of Participants Who Reported Positive Overall Efficacy and Tolerability at 24-hour Follow-up
Description: Patient's assessment of overall efficacy and tolerability was assessed by asking the question, "The next time you come to the emergency department with a headache or migraine, do you want to be given the same medication?". A "yes" response was considered positive assessment of overall efficacy and tolerability.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac, Intranasal | Ketorolac, Intravenous
Number analyzed (Participants) | 24 | 22
Participants | 19 | 21

9. Other Pre Specified Outcome: Number of Participants Who Reported Sustained Headache Freedom at 24-hour Follow-up
Description: Sustained headache freedom defined as achieving headache freedom (i.e. headache pain intensity of "none"), and maintaining this level for 24 hours without the use of rescue medications after emergency department discharge.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac, Intranasal | Ketorolac, Intravenous
Number analyzed (Participants) | 24 | 23
Participants | 7 | 12

10. Other Pre Specified Outcome: Number of Participants Who Reported Sustained Headache Relief at 24-hour Follow-up
Description: Sustained headache relief defined as achieving headache relief (i.e. headache pain intensity of "mild" or "none") and maintaining this level for 24 hours without the use of rescue medications after emergency department discharge.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac, Intranasal | Ketorolac, Intravenous
Number analyzed (Participants) | 24 | 23
Participants | 7 | 12

11. Other Pre Specified Outcome: Number of Participants Who Used Rescue Medication(s) Within 24 Hours After Emergency Department Discharge
Description: Rescue medications used after emergency department discharged defined as an analgesic taken by the participant at home to reduce pain associated with their headache.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac, Intranasal | Ketorolac, Intravenous
Number analyzed (Participants) | 18 | 19
Participants | 12 | 8

ADVERSE EVENTS:
Time Frame: 24 hours after discharge from emergency department.
Arm/Group | Ketorolac, Intranasal | Ketorolac, Intravenous
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/29
Other Adverse Events (participants affected / at risk) | 5/27 | 6/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketorolac, Intranasal (N=27) | Ketorolac, Intravenous (N=29)
Nausea (Gastrointestinal disorders) | 2 | 1
Dizziness (Nervous system disorders) | 1 | 1
Sleepiness (Nervous system disorders) | 0 | 1
Other (Nervous system disorders) | 2 | 3 — "Feeling cold", "less focus, feel off", transient extremity sensory complaints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT02358681/Prot_SAP_000.pdf